CLINICAL TRIAL: NCT03949556
Title: Internet-based Programmes for the Prevention of Suicidal Ideation in Medical Students
Acronym: InforMed
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: InforMed
Record Dates: First submitted 2019-05-13; First posted 2019-05-14 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: An open three-arm randomized controlled trial will be conducted to assess the effectiveness of two programmes of suicide prevention in fourth-year medical students and first-year interns; one based on stress management using cognitive and behavioural principles and the other on health promotion. Their respective effectiveness will be compared with a control condition. Participants will be assessed using validated questionnaires online at inclusion (before intervention) and at 6 (end of the intervention), 12, and 18 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention program - stress management program (Experimental): This intervention program on stress management is developed to prevent suicidal ideation in medical students and residents.
  Interventions: Other: Videos and/or SMS
- Intervention program - health promotion program (Active Comparator): This intervention program on health promotion is developed to prevent suicidal ideation in medical students and residents.
  Interventions: Other: Videos and/or SMS
- Control condition - general information (Placebo Comparator): Participants will receive weekly emails and SMSs, over the same periods of time, with general information about health except mental health, e.g. prevention of melanoma, dental care….
  Interventions: Other: Videos and/or SMS

INTERVENTIONS:
Other: Videos and/or SMS — Participants assigned to one of the intervention programmes will watch videos on a website for two months then will receive SMSs for four months.

SUMMARY:
Two programmes have been built to prevent suicidal ideation; one focuses on stress management based on cognitive and behavioural principles and the other on health promotion.

DETAILED DESCRIPTION:
The main objective will be assessing their respective effectiveness on suicidal ideation (at least one occurrence over a 12-month period after the end of the intervention), through a randomized controlled trial, in medical students and interns.

ELIGIBILITY:
Inclusion Criteria:

* Being registered in the fourth year of medical studies or in the first year of residency (internship), as they appear as two critical periods over medical studies
* Being registered in the i-Share cohort
* 18 year-old and over
* Speaking and reading French
* Having given an informed consent
* Ability to understand the type, the aims and the methodology of the study
* Agreement for online clinical assessment
* Having a mobile phone number and an e-mail address
* To be beneficiary of a health insurance programme

Exclusion Criteria:

* Refusing to participate
* Protective supervision: curatorship, guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2544 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation observed at least at one of the three assessment contacts (6, 12, 18 months). | 18 months
  The electronic Columbia-Suicide Severity Rating Scale (e-CSSRS) will be used to investigate suicide ideation & behaviors.
  Questionnaire was developped with NIMH support to screen & quantify suicide risk using consecutive questions. No score is computed when using this scale.
  Questionnaire investigates suicide ideation using several questions (response yes/no):
  1. Have you wish you were dead?
  2. Have you actually had any thought of killing yourself? If 1 and/or 2 are answered "yes", 4 other questions are asked. For this study, suicide ideation will be considered as a "yes" answered to question 1 or 2.

SECONDARY OUTCOMES:
Suicidal behaviour identified at least once after the intervention. | 18 months
  The electronic Columbia-Suicide Severity Rating Scale (e-CSSRS) will be used to investigate suicide ideation and behaviors.
  This questionnaire was developped with NIMH support to screen and quantify suicide risk using consecutive questions. No score is computed when using this scale.
  The questionnaire investigates also suicide behaviours using questions (response yes/no) on
  * actual attempt (have you made a suicide attempt? Have you done anything to harm yourself? have you done anything dangerous where you could have died?)
  * interrupted attempt
  * aborted or self-interrupted attempt
  * preparatory acts or behavior
  For the present study, suicide behavior will be considered as a "yes" to any of these 4 questions.

CONTACTS AND LOCATIONS:
Overall Officials: MARIE TOURNIER, MD, Prof, Principal Investigator — Centre Hospitalier CHARLES PERRENS
Locations (1):
- Centre Hospitalier Charles PERRENS, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No